CLINICAL TRIAL: NCT05969821
Title: National Cohort of Patients With Dysimmune Manifestations With or Without Clonal Hematopoiesis
Brief Title: Clonal Hematopoiesis of Immunological Significance
Acronym: CHIS
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Sorbonne University (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Club MINHEMON (MEDECINE INTERNE, HEMATO ET ONCO) (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP231600
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Immune System Diseases; Autoimmune Diseases; Inflammation; Autoinflammatory Diseases; Vexas Syndrome; Hematopoiesis Clonal; Clonal Hematopoiesis of Indeterminate Potential; Hematologic Diseases; Myelodysplastic-Myeloproliferative Diseases; Leukemia Myelomonocytic Chronic; Myelodysplastic Syndromes; Myeloproliferative Disorders; Lymphoproliferative Disorders; Lymphoma; Leukemia; Monoclonal Gammopathy of Undetermined Significance
Keywords: Inflammation; Autoinflammatory Diseases; Vexas syndrome; Autoimmune Diseases; Clonal Hematopoiesis of Indeterminate Potential; Myelodysplastic-Myeloproliferative Diseases; Lymphoproliferative Disorders; Monoclonal Gammopathy of Undetermined Significance
MeSH Terms: conditions — Immune System Diseases; Autoimmune Diseases; Inflammation; VEXAS syndrome; Hematologic Diseases; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myelomonocytic, Juvenile; Myelodysplastic Syndromes; Myeloproliferative Disorders; Lymphoproliferative Disorders; Lymphoma; Leukemia; Monoclonal Gammopathy of Undetermined Significance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Dysimmune manifestations with or without clonal hematopoiesis: Dysimmune manifestations with or without clonal hematopoiesis
  Interventions: Other: observational cohort study

INTERVENTIONS:
Other: observational cohort study — observational cohort study

SUMMARY:
Ambispective, national, multicenter observational cohort study aimed at characterizing the satellite dysimmune manifestations of clonal hematopoiesis, including Vexas (Vacuoles, E1 enzyme, X-linked, Autoinflammatory and Somatic) syndrome.

DETAILED DESCRIPTION:
The clinical spectrum of dysimmune manifestations associated with blood diseases is wide. The pathophysiology of these manifestations is not well understood and their management is poorly codified. This observational cohort aims to list the different clinical pictures, the therapeutic management and the prognosis of patients according to the type of dysimmune manifestations and the type of hemopathy. We wish to have an inventory of the demographic, genetic, clinical and evolutionary data of patients with an inflammatory manifestation associated or not with a myeloid or lymphoid hemopathy. This will make it possible to establish quantitative data on the morbidity and mortality of these rare diseases and to propose therapeutic trials for the most serious patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years old
* Confirmed dysimmune manifestations: clinical or biological abnormality or systemic disease
* Presence or absence of myeloid or lymphoid blood disease according to World Health Organization (WHO) classification

Exclusion Criteria:

* Persons benefiting from special protection: adults under guardianship and curatorship; people hospitalized without their consent and not protected by law; persons deprived of liberty.
* Persons not affiliated to the social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research concerns :
  * patients whose inflammatory disease without or with haemopathy is already known when the cohort is set up, and for whom data will be collected retrospectively and then prospectively
  * incident cases identified after the cohort was set up.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2045-09 (Estimated); Study Completion 2045-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of dysimmune manifestations associated with hematological disorders | Baseline
  Number of new cases

SECONDARY OUTCOMES:
VEXAS syndrome | 10 years
  Number of patients with VEXAS syndrome
Dysimmune manifestations other than VEXAS syndrome | 10 years
  Number of patients with dysimmune manifestations other than VEXAS syndrome
Myeloid hemopathy | 10 years
  Number of patients with myeloid hemopathy
Lymphoid hemopathy | 10 years
  Number of patients with lymphoid hemopathy
Clonal hematopoiesis of undeterminate potential | 10 years
  Number of patients with clonal hematopoiesis of undeterminate potential
Skin involvement | 10 years
  Number of patients with skin involvement
Musculoskeletal involvement | 10 years
  Number of patients with musculoskeletal involvement
Ocular involvement | 10 years
  Number of patients with ocular involvement
Vascular involvement | 10 years
  Number of patients with vascular involvement
Neurological involvement | 10 years
  Number of patients with neurological involvement
Digestive system involvement | 10 years
  Number of patients with digestive system involvement
Cardiac involvement | 10 years
  Number of patients with cardiac involvement
Pulmonary involvement | 10 years
  Number of patients with pulmonary involvement
Renal involvement | 10 years
  Number of patients with renal involvement
Therapeutic interventions received | 10 years
  Type and duration of therapeutic interventions received
Progression to acute myeloid leukemia | 10 years
  Number of patients who progressed to acute myeloid leukemia
Overall mortality | 10 years
  Overall mortality rate from all causes

CONTACTS AND LOCATIONS:
Overall Officials: Arsene MEKINIAN, MD PhD, Principal Investigator — Service de médecine interne, Hôpital Saint Antoine, APHP, Paris

IPD SHARING:
Plan to Share IPD: No